CLINICAL TRIAL: NCT07337837
Title: Immediate Implant Placement in Type ii Socket by Vestibular Socket Therapy Using Collagen Membrane (Randomized Controlled Clinical Trial)
Brief Title: Immediate Implant Placement in Type ii Socket by Vestibular Socket Therapy Using Collagen Membrane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0809-12/2023
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Immediate Implant; Vestibular Socket Therapy; Type II Socket

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental)
  Interventions: Procedure: vestibular socket therapy
- Control Group (Active Comparator)
  Interventions: Procedure: open flap surgery

INTERVENTIONS:
Procedure: vestibular socket therapy — patients will undergo immediate implant placement and a mucoperiosteal tunnel will be made through a vestibular incision till labial orifice of the socket, a collagen membrane will be inserted under the tunnel and stabilized by membrane tacks. The space between the membrane and implant will be filled with mixture of allograft and xenograft bone material and any autogenous bone chips harvested from local surgical sites.
  Arms: Study group
Procedure: open flap surgery — patients will undergo immediate implant placement combined with open flap surgery and labial plate augmentation.
  Arms: Control Group

SUMMARY:
Background: Immediate implant placement has become a routine and regular clinical practice. When the labial bone plate develops a dehiscence-type defect, delayed implant placement was recommended to give suitable amount of time for soft tissue thickening. However, it has a number of drawbacks, including a lengthy treatment period, the requirement for two surgical procedures, and a potential loss of facial contour. When immediate implant is placed with flap elevation and guided bone regeneration in type II socket, labial bone augmentation results were satisfactory, but in terms of soft tissue, it led to midfacial recession and loss of soft tissue contour, resulting in a compromised final esthetic result. To reduce these drawbacks, implant can be immediately placed by vestibular socket therapy using collagen membrane.

Aim of this study: To compare labial bone augmentation in immediate implant placement in type II extraction sockets by using collagen membrane placed by two different modalities.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with a single maxillary tooth (second bicuspid to second bicuspid) indicate for extraction due to fracture, badly decayed or endodontic lesionswith expected labial bone defect

Exclusion Criteria:

* Pregnancy.
* Patients with any systematic disease that could complicate the surgical phase or affect osseointegration as osteoporosis and uncontrolled diabetes mellitus.
* Periodontal disease or gingival recession.
* Heavy smokers (more than 30 cigarette / day).
* Patients with poor oral hygiene

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
change in buccal bone thickness | baseline, 3 months, and 6 months
  CBCT will be taken for each patient and Labial bone thickness means the distance between the implant surface and the outer surface of bone
change in buccal bone height | Baseline, 3 months, and 6 months
  Labial bone height means the distance between the apical end of the implant (which is projected on the baseline image) and the crest of the labial bone of both images

SECONDARY OUTCOMES:
Volumetric change of buccal soft tissue contour | Baseline and 6 months
  The impressions will be taken using lab scanner to create digital surface models in Standard Triangle Language (STL) format, all STL files will be imported to a digital software. The best-fit algorithm will be used to superimpose digital surface models, when comparing each area of interest (AOI) throughout out the follow-up period.
change in gingival esthetics | Baseline and 6 months
  The score incorporates seven domains: mesial papilla, distal papilla, soft tissue level, soft tissue contour, deficient alveolar process, soft tissue color, and texture. Each variable is scored from 0 to 2, with 2 being the best outcome. The total pink esthetic score will be calculated by adding the scores of the seven domains and ranged from 0 to 14 (best overall esthetic outcome).
chang in Modified Sulcus Bleeding Index | Baseline and 6 months
  a score of 0-3 will be assigned to each labial and palatal surface of the implant then the average for each implant will be calculated according to the following criteria: Score 0: No bleeding when a periodontal probe is passed along the gingival margin adjacent to the implant.
  Score 1: Isolated bleeding spots visible. Score 2: Blood forms a confluent red line on margin. Score 3: Heavy or profuse bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Alexandria, Egypt